CLINICAL TRIAL: NCT04573985
Title: Impact of the Eurékoi Serious Game on Family Caregivers of Patients With a Major Neurocognitive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-AOI-09
Record Dates: First submitted 2020-09-22; First posted 2020-10-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Family Caregiver of Patient With Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious Game Eurekoi intervention (Experimental): 1 session in group using the serious game eurekoi
  Interventions: Behavioral: Serious game Eurekoi intervention
- Control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Serious game Eurekoi intervention — 1 session in group using the serious game eurekoi
  Arms: Serious Game Eurekoi intervention

SUMMARY:
This study aims to assess the effectiveness of serious EUREKOI gambling on the anxiety of family caregivers of patients with newly diagnosed Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years old;
* Primary caregiver of a patient with a mild-stage major neurocognitive disorder newly diagnosed according to the DSM 5 criteria;
* Signature of informed consent.

Exclusion Criteria:

* Subject not speaking French, not reading French
* Subject with visual impairment
* Subject under tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Efficacity of the serious game Eurekoi on anxiety of familial caregiver of patient with Alzheimer Disease | 3 months
  Auto-evaluation of anxiety using Spielberger inventory (score between 20 and 80 ; the higher the score, the greater the anxiety)

SECONDARY OUTCOMES:
Change of knowledge of familial caregiver about cognitive troubles | 3 months
  Multiple choice questionary
Evaluate satisfaction of the familial caregivers about the session with the game EUREKOI | 3 months
  questionary of satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France